CLINICAL TRIAL: NCT04446988
Title: Ultrasound Versus Fluoroscopic Guided Sacroiliac Joint Injection In Patients With Chronic Sacroiliac Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, DR. Abd El-Raheem Mahmoud, Clinical Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14102019
Record Dates: First submitted 2020-05-19; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Sacro-Iliac Spondylosis
Keywords: Sacroiliac

STUDY DESIGN:
Intervention Model Description: Sacroiliac joint injection with local anesthetic and steroid using ultrasound Versus fluoroscopy in sacroiliitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound(US) (Experimental): Sacroiliac joint injection using ultrasound
  Interventions: Device: Sacroiliac joint injection
- Fluoroscopy(FL) (Experimental): Sacroiliac joint injection using fluoroscopy
  Interventions: Device: Sacroiliac joint injection

INTERVENTIONS:
Device: Sacroiliac joint injection — Injection of sacroiliac joint with local anesthetic and steroid

SUMMARY:
Sacroiliac joint injection in sacroiliitis

DETAILED DESCRIPTION:
Comparison of ultrasound guided and fluoroscopic guided sacroiliac joint injection

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sacroiliitis.
* At least 3 positive physical examination maneuvers [FABER (flexion, abduction, and external rotation), POSH (posterior shear), REAB (resisted abduction), Fortin's finger test],
* Moderate to severe pain (NRS pain score ≥ 3/10) refractory to oral anti-inflammatory.
* Age from 18ys to 60ys.

Exclusion Criteria:

* Ages less than 18 or more than 85 years.
* Body Mass Index (BMI) above 35 kg/m2.
* A diagnosis of severe anxiety or depression and other psychological disorders.
* Allergy to local anesthetics or steroids and pregnancy.
* Multiple comorbidities (renal , hepatic, cardiac).
* Coagulation disorder as bleeding tendency and platelet dysfunction.
* Contraindication for prone position or radiological exposure.
* Patient refuse .
* Pain suggestive of bilateral sacroiliac joint involvement (it would have been difficult to assess pain and disability secondary to each SIJ).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) pain scores | 3 months
  It measures pain intensity (0 no pain - 10 worst pain imaginable)
Oswestry disability index score | 1 month
  It evaluates the physical function (0% minimal disability - 100% bed - bound patient)

SECONDARY OUTCOMES:
Analgesic requirement | 1 month
  It shows if the patient needs analgesic or not compared to pretreatment (type and dose in mg)
Patient satisfaction ( global perceived effect on a 7-point scale (GPE) ) | 3 months
  It shows if the patient satisfied with the procedure or not (1= worst ever - 7= best ever)
Procedure time | Procedure
  It measures the seconds of procedure in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ka Mickhael, Ass. pr., Principal Investigator — Minia University
Locations (1):
- ASSIUT University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benson DA, Cavanaugh M, Clark K, Karsch-Mizrachi I, Lipman DJ, Ostell J, Sayers EW. GenBank. Nucleic Acids Res. 2013 Jan;41(Database issue):D36-42. doi: 10.1093/nar/gks1195. Epub 2012 Nov 27. PMID 23193287